CLINICAL TRIAL: NCT06078891
Title: Does BCG Vaccination Reduce Biomarkers of Alzheimer's Disease?
Acronym: BCG-AD
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tamir Ben-Hur (Other)
Collaborators: Hebrew University of Jerusalem (Other)
Responsible Party: Sponsor-Investigator, Tamir Ben-Hur, Professor and Chair, The Brain Divison, Hadassah Medical Organization
Organization: Hadassah Medical Organization (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BCG-AD HMO-CTIL
Record Dates: First submitted 2023-08-06; First posted 2023-10-12 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Alzheimer Disease, Late Onset
MeSH Terms: conditions — Alzheimer Disease | interventions — BCG Vaccine

STUDY DESIGN:
Intervention Model Description: A single group in treated patients to follow changes in plasma biomarkers levels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BCG vaccinated patients (Experimental): A single arm experiment to examine the effect of 3 standard intradermal vaccinations with BCG (at times 0, 1 month and 12 months) on plasma biomarkers.
  Interventions: Biological: BCG vaccine

INTERVENTIONS:
Biological: BCG vaccine — Three intra-dermal vaccinations over a period of one year.

SUMMARY:
The goal of this clinical trial is to test whether vaccination with the BCG vaccine may improve the blood level of a biomarker of Alzheimer's disease (AD) in participants who are cognitively- and functionally- intact elderly (70-80 years old) participants, who display pathologically high levels of the blood biomarker.

The main questions it aims to answer are:

* Does BCG vaccination lower the plasma level of phosphorylated Tau protein (p-tau181).
* Do vaccinated participants remains stable cognitively.

Participants will be asked to:

* Undergo cognitive and behavioral evaluation.
* Receive 3 BCG vaccinations over the course of 1 year.
* Perform blood tests on several occasions. All participants will be treated and followed.

DETAILED DESCRIPTION:
Brain accumulation of insoluble Beta-Amyloid and of hyperphosphorylated tau protein -rich neurofibrillary tangles in Alzheimer's disease (AD), accompanied by oxidative stress and sustained inflammation develops approximately 20 years before appearance of symptomatic dementia. These years should be regarded as an incubation period of a deadly condition during which early therapeutic intervention may increase the likelihood of obtaining a significant disease modifying effect. Early diagnosis at the pre-symptomatic stage has been hindered by the lack of reliable, inexpensive and non-invasive biomarkers of disease. Recent developments have enabled the measurement of plasma p-tau181 level, which has almost 90% sensitivity and specificity for diagnosing AD. As these biomarkers identify AD pathology prior to clinical presentation, they enable identifying pre-symptomatic patients, with potential of early intervention. P-tau181, neurofilament light (NfL) and GFAP biomarkers may also serve as outcome measures, corresponding to the severity of active neurodegenerative disease in AD.

The investigators propose to select 60 individuals who are at high risk for developing AD dementia for a single-arm prospective intervention study, by screening cognitively- and functionally-intact elderly population with non-genetic AD risk factors (around 250 individuals, 70-79 years old) for high plasma p-tau181 level. The current lack of any disease modifying drug in AD urged them to test if BCG vaccination can prevent, or at least postpone AD. The rationale is based on multiple scientific observations and on the dramatic reduction (by 30-50%) in development of dementia in elderly patients with bladder cancer who were treated with multiple intra-vesicular BCG instillations. Accumulating data argue for the critical role of the immune system in the course of AD. BCG through its immune-modulation properties (Tregs, pDCs and IL10 enhancement, M1:M2 macrophage balance) may mitigate the inflammatory process component of AD and therefore may prevent or delay full blown AD.

In this single arm prospective study, three BCG vaccinations will be provided to the 60 recruited participants over one year. At recruitment and at three times during the two years' study period, they will be tested for plasma p-tau181 level, and for plasma Nfl and/or GFAP using SIMOA technology. The baseline p-tau181 will serve as a reference value for monitoring individual response to the BCG vaccinations during the study, as well as the group trend for the total Tau biomarker. The investigators will also study the effect of BCG vaccination on the dynamics of the cognitive performance of the selected individuals.

The investigators hypothesize that BCG vaccination in individuals with high-risk pre-symptomatic Alzheimer's disease will reduce active brain disease, as determined by blood biomarkers' levels and will mitigate cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* 70-80 years old patients with self-reported preserved cognitive function and instrumental activities of daily life (iADL).
* MoCA score of ≥26.
* Increased plasma p-tau181 level.

Exclusion Criteria:

* Extrapyramidal signs, documented CVA, existence of multi-infarct dementia or fronto-temporal dementia according to clinical impression by treating cognitive neurologist.
* Active cancer, severe cardio-pulmonary disease or other medical condition which negatively affects ability to evaluate patients and complete follow-up.
* Active glucocorticoids treatment, chronic immunosuppressive medications, or currently living with an immunosuppressed individual to prevent an adverse event from the administration of this live vaccine.
* Above 10mm induration diameter at 48 hours after initial PPD test.
* Inability to sign an informed consent due to psychiatric or dementing condition.

Ages: 70 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Plasma phosphorylated Tau (p-tau181) biomarker level, measured in picogram/ml by SIMOA technology. | 1.5 years
  Four measurements of plasma p-tau181 levels (range 1-100 picogram/ml)

SECONDARY OUTCOMES:
Cognitive deterioration by Montreal Cognitive Assessment (MoCA) test | 1.5 years
  Cognitive evaluation by MoCA test (score 0-30) at recruitment and after 1.5 years
Plasma neurofilament-light levels by SIMOA technology | 1.5 years
  Two measurements of neurofilament-light levels (range 1-100 picogram/ml) by SIMOA technology

CONTACTS AND LOCATIONS:
Overall Officials: Tamir Ben Hur, MD PhD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Department of Neurology, Hadassah medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No